CLINICAL TRIAL: NCT02830256
Title: Psychometric Measurements of Three Nociception Assessments Methods in Intubated Brain Injured Critical Care Patients
Acronym: D co réa
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9673; 2016-A00748-43 (Other: RCB number)
Record Dates: First submitted 2016-06-13; First posted 2016-07-12 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2017-04

CONDITIONS: Intubated Brain Injured
Keywords: Intensive care unit; Neuro-ICU; Pain; Intubation; critical care; patients
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: NCS-I (Nociception Coma Scale adapted intubated patients) — Every included patient will be assessed by the 3 methods 3 times (before, during, after the procedure fo care) in 3 conditions. There will be 2 painful conditions usually performed in ICU (Nursing and bronchoaspiration) and a painless condition (RASS assessment).

SUMMARY:
Nociception in intensive care unit is frequently evaluated with some tools such as BPS (Behavioral Pain scale) and NCS (Nociception coma scale). These scales were not validated in intubated and brain injured ICU patients. The investigators propose to validate the NCS adapted for intubated patients (NCS-I) in comparison with the recommended scale (BPS) and the Pupillary response (videopupillometry) to noxious stimulation (common procedure of care).

DETAILED DESCRIPTION:
Nociception in intensive care unit is frequently evaluated with some tools such as BPS (Behavioral Pain scale) and NCS (Nociception coma scale). These scales were not validated in intubated and brain injured ICU patients. The investigators propose to validate the NCS adapted for intubated patients (NCS-I) in comparison with the recommended scale (BPS) and the Pupillary response (videopupillometry) to noxious stimulation (common procedure of care).

ELIGIBILITY:
Inclusion criteria:

* Adult, > or equal to 18-yr
* Admission to intensive care unit
* Brain injured and intubated patient
* Signs of awakening after the interruption of sedation
* Impossibility to self-report pain intensity

Exclusion criteria:

* Eye injuries (glaucoma, keratitis, conjunctivis, cataract)
* Neurodegenerative attack
* Brainstem damage
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admission to intensive care unit
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Difference in pain scores or pupillary diameter measures at rest and during care procedures | Through study completion (30 months)
  Discriminant validity between NCS-I, BPS and pupillary measurements will follow current recommended method for psychometric assessment of pain tools in critical care patients (Pain Agitation and Delirium Guidelines from the Society of Critical Care Medicine, Barr et al. Crit Care Med 2013). Mann-Whitney-Wilcoxon test will be used to compare values obtained at rest and during the procedures of care.

SECONDARY OUTCOMES:
Weight kappa coefficient for pain using the NCS-I | Through study completion (30 months)
  Reliability of NCS-I and BPS will follow current recommended method for psychometric assessment of pain tools in critical care patients (Pain Agitation and Delirium Guidelines from the Society of Critical Care Medicine, Barr et al. Crit Care Med 2013).
Weight kappa coefficient for pain using the BPS | Through study completion (30 months)
  Weighted kappa coefficient will be used to measure inter-observers agreement using the two subjective pain scales (NCS-I and BPS).

CONTACTS AND LOCATIONS:
Overall Officials: GERALD CHANQUES, MD PH D, Study Director — University Hospital, Montpellier; Pierre François PERRIGAULT, MD, Study Chair — University Hospital, Montpellier; Christine BERNARD, CRNA, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernard C, Delmas V, Duflos C, Molinari N, Garnier O, Chalard K, Jaber S, Perrigault PF, Chanques G. Assessing pain in critically ill brain-injured patients: a psychometric comparison of 3 pain scales and videopupillometry. Pain. 2019 Nov;160(11):2535-2543. doi: 10.1097/j.pain.0000000000001637. PMID 31188267